CLINICAL TRIAL: NCT06335667
Title: Outcomes With Multi Parametric MRI (mpMRI) Compared to Diagnostic Transurethral Resection of Bladder Tumor (TURBT) in Patients With Suspected Muscle-Invasive Bladder Cancer - a Pilot Study
Brief Title: mpMRI Compared to Diagnostic TURBT in Patients With Suspected Muscle-Invasive Bladder Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Nataliya Mar, Associate Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4565; UCI 23-72 (Other: UCI CFCCC)
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Urothelial Bladder Cancer; Muscle-Invasive Bladder Cancer
Keywords: mpMRI; TURBT; VI-RADS score
MeSH Terms: interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- mpMRI + Diagnostic TURBT (Experimental)
  Interventions: Diagnostic Test: mpMRI + Diagnostic TURBT

INTERVENTIONS:
Diagnostic Test: mpMRI + Diagnostic TURBT — mpMRI in addition to the TURBT surgical procedure

SUMMARY:
This is a pilot, single arm, prospective study that aims to validate the accuracy of the VI-RADS score obtained via multi-parametric magnetic resonance imaging (mpMRI) compared to pathologic cancer stage obtained via diagnostic transurethral bladder tumor resection (TURBT) as well as compare the clinical and quality of life outcomes between these diagnostic modalities in patients with suspected muscle-invasive bladder cancer (MIBC).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or greater at the time of consent.
* Suspected muscle-invasive bladder cancer by tumor appearance on initial routine cystoscopy as determined by the UCI-affiliated urologist performing this procedure.
* ECOG Performance Status of 0-3.
* Patients must have the ability to understand and the willingness to sign a written informed consent document (prior to the initiation of the study and any study procedures).
* Patients must be willing and able to comply with the scheduled visits, imaging plan, follow up plan, and other specified study procedures in the opinion of the Investigator.

Exclusion Criteria:

* Prior TURBT within 120 days of study entry.
* Prior therapy for bladder cancer within 120 days of study entry.
* Inability to tolerate mpMRI or associated contrast.
* Inability to tolerate TURBT or associated anesthesia.
* ECOG Performance Status of 4.
* Female patient who is known to be pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of concordance between VI-RADS score of 4 or 5 (i.e. muscular propria is likely or very likely) on mpMRI and pathologic muscularis propria invasion (i.e. pT2 tumor stage) on diagnostic TURBT. | Up to 1 year
  VI-RADS is a five-point scoring system developed to standardize imaging and reporting of bladder tumor invasiveness on mpMRI. It predicts the degree of possible muscular propria invasion ("muscle-invasiveness") of bladder tumors. Once diagnostic TURBT is performed, the VI-RADS score from mpMRI will be compared to the pathologic tumor (T) stage from a diagnostic TURBT to assess for concordance.

SECONDARY OUTCOMES:
Progression free survival (PFS) with mpMRI compared to diagnostic TURBT | up to 5 years
  Time from diagnostic test to cancer progression, recurrence, or death.
Time from intervention that determines invasiveness of bladder tumors (i.e. diagnostic TURBT versus mpMRI) to initiation of cancer-directed therapy | up to 5 years
Time from initial cystoscopy to intervention that determines invasiveness of bladder tumors (i.e diagnostic TURBT versus mpMRI). | up to 5 years
Incidence of adverse events with mpMRI versus diagnostic TURBT. | up to 5 years
Patient Quality of Life with mpMRI versus diagnostic TURBT. | up to 5 years
  As assessed by quality of life questionnaires
Incidence of repeat TURBT. | up to 5 years
Diagnostic healthcare expenditure with mpMRI versus diagnostic TURBT | up to 5 years
  in dollars

CONTACTS AND LOCATIONS:
Overall Officials: Nataliya Mar, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center University of California, Irvine, Orange, California, United States